CLINICAL TRIAL: NCT02295371
Title: Medication Incidents in Primary Care Medicine: A Study by the Swiss Federal Sentinel Reporting System
Brief Title: Medication Incidents in Primary Care Medicine
Acronym: MIPC
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Sponsor
Other Study IDs: MIPC
Record Dates: First submitted 2014-11-10; First posted 2014-11-20 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Medication Incidents
Keywords: Drug therapy; Patient safety; Polydrug therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with an incident: Patients undergoing a safety incident while being treated with drugs

SUMMARY:
Prospective reporting of safety incidents concerning drug treatment by approximately 120 primary care physicians or pediatricians during 2015.

DETAILED DESCRIPTION:
Objectives: Patient safety is a major concern in healthcare systems worldwide. Although most safety research has been conducted in the inpatient setting, evidence indicates that medical errors and adverse events pose a serious threat for patients in the primary care setting as well, since most patients receive ambulatory care. Information about frequency and outcomes of safety incidents in primary care is required to identify risks or "hot spots," to prioritize them and to take the action as needed.

Methods:

Participants: Patients undergoing drug treatment by approximately 120 primary care physicians or pediatricians reporting to the Sentinel system.

Collection of data: Questionnaires for cases, for clinical denominator data, and for physician practice specification.

Study intervention: none.

Primary outcome:

● To describe the type, frequency, seasonal and regional distribution of medication incidents

Secondary outcomes:

● To elucidate risk factors like age, gender, poly-medication, morbidity, foreign care, hospitalization.

Statistics: Descriptive statistics, logistic regression. Estimated sample size: 500.

Flow chart: January 2015: Baseline physicians questionnaire. May 2015: Denominator data collection during 14 d. December 2015: Final physicians questionnaire. January to December 2015: Collection of case questionnaires / Counting of daily patient-to-physician contacts. After December 2015: Statistical Evaluation of data, publication.

ELIGIBILITY:
Inclusion Criteria:

* Any erroneous event (as defined by the physician) related to the medication process interfering with normal treatment course

Exclusion Criteria:

* Lacking treatment effect, adverse drug reactions or drug-drug or drug-disease interactions, without detectable treatment error.
* Refusal of patients to refer data to the Sentinel system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients consulting primary care practices
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
type, frequency, seasonal and regional distribution of medication incidents | 12 monthes
  Descriptives

SECONDARY OUTCOMES:
possible risk factors for medication incidents like age, gender, poly-medication, morbidity, previous hospitalization | 12 monthes
  Logistic regression

CONTACTS AND LOCATIONS:
Overall Officials: Markus P. Gnädinger, MD, Principal Investigator — Institute for General Medicine, Zurich University Hospital
Locations (1):
- Praxis Dr. med. Markus Gnaedinger, Steinach, Canton of St. Gallen, Switzerland

REFERENCES:
- [Derived] Gnadinger M, Herzig L, Ceschi A, Conen D, Staehelin A, Zoller M, Puhan MA. Chronic conditions and multimorbidity in a primary care population: a study in the Swiss Sentinel Surveillance Network (Sentinella). Int J Public Health. 2018 Dec;63(9):1017-1026. doi: 10.1007/s00038-018-1114-6. Epub 2018 May 21. PMID 29786762
- [Derived] Gnadinger M, Ceschi A, Conen D, Herzig L, Puhan M, Staehelin A, Zoller M. Medication incidents in primary care medicine: protocol of a study by the Swiss Federal Sentinel Reporting System. BMJ Open. 2015 Apr 23;5(4):e007773. doi: 10.1136/bmjopen-2015-007773. PMID 25908679